CLINICAL TRIAL: NCT00318994
Title: Evaluation of Pancreatic Tissue Penetration of Meronem® in the Prophylaxis of Septic Complications in Severe Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3591/9010; D9211C09010
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Meropenem

INTERVENTIONS:
Drug: Meropenem

SUMMARY:
To measure meropenem pancreatic tissue penetration in subjects with severe pancreatitis requiring surgery between 30 to 60 minutes after a bolus of 1 g IV meropenem given during the induction period of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of severe pancreatitis requiring surgery according to the protocol of each Institution.
* Informed consent signed by the subject
* Subjects who have received prophylactic antibiotics for previous invasive procedures different from surgery may be included

Exclusion Criteria:

* Will of the subject not to be included
* Subjects who have not signed the informed consent
* Subjects with known hypersensibility to carbapenems, penicillins, or cephalosporins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6
Dates: Start 2002-02; Primary Completion 2005-09 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To measure meropenem pancreatic tissue penetration in subjects with severe pancreatitis requiring surgery between 30 and 60 minutes after a bolus of 1 g IV meropenem applied during induction of anesthesia.

SECONDARY OUTCOMES:
To describe the incidence of infectious complications during the first 30 days after surgery in subjects with severe pancreatitis receiving IV meropenem at a dose of 1 g every 8 hours during 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Columbia Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Bogotá, Colombia